CLINICAL TRIAL: NCT02434913
Title: HUD: Proximal Interphalangeal (PIP) Joint Implant Finger Prosthesis
Brief Title: HUD: PIP Joint Implant
Status: No longer available | Type: Expanded Access
Sponsor: The Hawkins Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00026976
Record Dates: First submitted 2014-09-15; First posted 2015-05-06 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Arthrosis; Osteoarthrosis
Keywords: Proximal interphalangeal joint deformity; Arthroplasty
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Device: SR PIP Implant System — HUD for use in arthroplasty of the PIP joint

SUMMARY:
This surgery involves the use of a finger joint replacement device for treatment of patients with certain kinds of arthritis (osteo - arthritis or post traumatic arthritis) and who expect to place their hands in heavy loading situations, or patients needing revision of a failed implant placed in the PIP joint. A joint replacement surgery is an operation where the arthritic joint is removed and a metal and plastic joint is inserted to replace the natural joint. The surgery is expected to last about 2 hours. The procedure is done in the operating room and requires general anesthesia or an axillary block. (General anesthesia affects the entire body and is accompanied by a loss of consciousness. An axillary block results in anesthesia of the hand and forearm only. A tourniquet is applied to the arm to prevent bleeding during the surgery.)

ELIGIBILITY:
Inclusion Criteria:

* Patients with disability of the their finger from arthrosis

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Allen, MD, Principal Investigator — Steadman Hawkins Clinic of the Carolinas - Greenville Health System